CLINICAL TRIAL: NCT02160561
Title: Feasibility of Upright Bed Position in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00023156
Record Dates: First submitted 2014-05-27; First posted 2014-06-10 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness; Acute Respiratory Failure; Adult Syndrome
Keywords: mechanical; ventilation; acute; respiratory; failure
MeSH Terms: conditions — Critical Illness; Propping Zerres syndrome; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Experimental - Intervention Arm patients who are in critical illness with acute respiratory failure and are mechanically ventilated will be placed in an upright reverse trendelenburg position
  Interventions: Other: Intervention Arm

INTERVENTIONS:
Other: Intervention Arm — Placing patients who are in critical illness with acute respiratory failure and are mechanically ventilated in an upright reverse trendelenburg position

SUMMARY:
Lower lobe atelectasis of the lung is common in Acute Respiratory Distress Syndrome (ARDS) and has the potential to adversely impact lung compliance and intra-pulmonary shunt. The cephalic shift of the diaphragm and dorsal atelectasis associated with the commonly used supine position might also contribute to this shunt. Reports indicate that obese patients may be more likely to develop dorsal atelectasis than non-obese patients.

The investigators hypothesized that opening the body position angle at the waist from a typical head of bed at 30 degrees to one similar to a more upright reverse trendelenburg position, would alter the position of the diaphragm downward, allowing for improved aeration of lung bases. Thus, the investigators examined the upright body positioning in mechanically ventilated patients with ARDS primarily by evaluating for effects on oxyhemoglobin saturation (O2sat), Tidal Volume (TV) and Respiratory Rate (RR).

DETAILED DESCRIPTION:
Acute respiratory failure and acute respiratory distress syndrome is a life-threatening occurrence. The annual incidence of ARDS is 141,500 patients, with 59,000 deaths, and a cost of 1,642,000 hospital days/year. Within this population, special care needs of obese patients are becoming a clinically important entity within the Intensive Care Unit (ICU). ICU literature on body positioning for obese mechanically ventilated patients is limited. Currently, intubated obese patients are placed in the supine position with the head of bed elevated at 30 degrees. The 30 degree head up position has been adopted for all patients as a reflection of the Ventilator Associated Pneumonia prevention literature. In all critically ill patients on mechanical ventilation, a cephalic shift of the diaphragm along with dorsal atelectasis of the lung occurs. In obese patients this alteration may be associated with greater degree of impairment in lung compliance and gas exchange as compared to non-obese ventilated patients. It is possible that current ICU body positioning recommendations for obese mechanically ventilated patients may be detrimental due to the obese abdominal compartment hampering normal diaphragm function and position.

In supine, intubated, mechanically ventilated patients it has long been noted that lower lung lobes become atelectatic soon after intubation due to several factors such as accumulation of fluids, air closure, and a cephalic shift of the diaphragm. Obese patients develop more atelectasis during anesthesia than non-obese patients. There have been attempts to correct this iatrogenic complication in critically ill patients such as placement of patients in the prone position. Prone positioning does resolve the dorsal atelectasis and shows improvement in hypoxia. However there is no mortality benefit with prone positioning. Also, continuous lateral rotational patient positioning on mechanical ventilation has shown similar effects7. Specific literature with regards to obese patients and their unique susceptibility towards this phenomenon is limited.

As BMI increases there is an associated reduction of lung volumes, expiatory reserve volume, and functional reserve capacity. It is also known that in the reverse trendelenburg position, there is a gravitational pull allowing abdominal contents to descent toward the pelvis. This position of the abdominal contents allows for a more functional diaphragm position. One observational study 10 conducted a 12 hour intervention which examined upright position with patients' body in a straight line at 40-45 degrees (i.e., reverse trendelenburg-no bend at the waist). This study demonstrated a significant increase in the PaO2/FiO2 ratio (ie, oxygenation) during upright position.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Chest radiograph must show parenchymal lung infiltrates.
* Acute Lung Injury
* Study shall occur 96 hours after consent has been obtained

Exclusion Criteria:

* Hemodynamic instability and/or use of a vasopressor within the last 6 hours prior to enrollment.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with change in hemodynamic stability from baseline when placed in upright position | Three hours
  Hemodynamic stability will be determined by changes from baseline in blood pressure or heart rate when participants are placed in an upright position.

SECONDARY OUTCOMES:
Number of participants with change in Oxyhemoglobin Saturation from baseline when placed in upright position | Three hours
  Oxyhemoglobin saturation levels will be monitored when participant is placed in upright position. Change from baseline level will be recorded.
Number of participants with Change in Tidal Volume from baseline when placed in upright position | Three hours
  Tidal volume will be monitored when participant is placed in upright position. Change from baseline level will be recorded.
Number of participants with change from baseline in Respiratory Rate when placed in upright position | Three hours
  Respiratory stability will be determined by changes from baseline in respiratory rate when participants are placed in an upright position.

OTHER OUTCOMES:
Number of participants with change from baseline in respiratory system compliance when placed in upright position | Three hours
  Respiratory System Compliance will be determined by changes from baseline in anxiety level and ventilation requirements when participants are placed in an upright position. Participants will be continually monitored and observed to note changes in anxiety on a comfort scale as well as any mechanical ventilator changes to mode, rate, and delivered oxygen percents required for comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Morris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Medical Intensive Care Unit, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strandberg A, Tokics L, Brismar B, Lundquist H, Hedenstierna G. Constitutional factors promoting development of atelectasis during anaesthesia. Acta Anaesthesiol Scand. 1987 Jan;31(1):21-4. doi: 10.1111/j.1399-6576.1987.tb02513.x. PMID 3825472